CLINICAL TRIAL: NCT05963191
Title: Evaluation of the CAD-EYE System for the Detection of Colorectal Neoplastic Lesions in Patients With Lynch Syndrome
Brief Title: CAD-EYE System for the Detection of Neoplastic Lesions in Patients With Lynch Syndrome
Acronym: CADLYNCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PERROD Guillaume (Other)
Responsible Party: Sponsor-Investigator, PERROD Guillaume, Principal Investigator, Medical Doctor, French Society of Digestive Endoscopy
Organization: French Society of Digestive Endoscopy (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SFED 156
Record Dates: First submitted 2023-07-10; First posted 2023-07-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Lynch Syndrome
Keywords: Lynch Syndrome; CAD EYE; adenoma detection rate; colorectal screening; artificial intelligence
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD-EYE group: Colorectal cancer screening with CAD EYE colonoscopy (Experimental): The colonoscopy procedure for each patient will be no different from a conventional colonoscopy examination. In the CAD EYE group, descent is performed under white light, with the CAD EYE system switched on (device with CE mark). When polyps are detected, they are rigorously described and histological predictions of endoscopist and CAD EYE will be reported separately.
  Interventions: Device: Colorectal cancer screening with CAD EYE colonoscopy
- CE group : Colorectal cancer screening with indigo carmine chromo colonoscopy (No Intervention): The colonoscopy procedure for each patient will be no different from a conventional colonoscopy examination. In the CE group, descent is performed under white light with indigo carmin chromoendoscopy (0.4%) applied through a catheter spray. When polyps are detected, they are rigorously described and histological prediction of the endoscopist reported.

INTERVENTIONS:
Device: Colorectal cancer screening with CAD EYE colonoscopy — The colonoscopy procedure for each patient will be no different from a conventional colonoscopy examination. A colonoscopy is considered complete if the endoscope reaches the appendicular orifice or the terminal ileum. In line with recommendations, water lavage (using a lavage pump) and aspiration of food residues will be performed on ascent and/or descent to visualize the entire colonic mucosa.
  In the CAD EYE group, descent is performed under white light, with the CAD EYE system switched on. When polyps are detected, they are rigorously described and histological predictions of endoscopist and CAD EYE will be reported separately. Then polyps will be removed by polypectomy or mucosectomy. Removed polyps are then sent for anatomopathological analysis.
  Arms: CAD-EYE group: Colorectal cancer screening with CAD EYE colonoscopy

SUMMARY:
Lynch syndrome (LS) is the most common genetic predisposition syndrome for colorectal cancer (CRC), responsible for around 2-4% of cancers. It is characterized by a pathogenic germline mutation in one of the DNA mismatch repair genes (path_MMR) MLH1, MSH2, MSH6, PMS2 or a deletion in the 3' region of the Epcam gene. Patients followed up for LS are at high risk of developing CRC at an early age, and have a high cumulative CRC risk. In this context, CRC screening by colonoscopy is of major importance, as it is associated with a reduction in both CRC incidence and mortality.

In France, the Institut National du Cancer (INCa) recommends colonoscopy with indigo carmine chromoendoscopy (CE), as it is associated with a significant increase in the adenoma detection rate (ADR) compared with white light. However, EC is not routinely performed in clinical practice, as it is a time-consuming technique requiring a dedicated slot with a trained operator.

Recent years have seen the emergence of artificial intelligence techniques for real-time polyp detection aids or CADe devices. These easy-to-use systems have shown very promising results compared with high-definition (HD) white light. Indeed, data from the first meta-analysis of 5 randomized controlled trials (4354 patients) confirmed a significantly higher ADD in the CADe group than in the HD group (36.6% vs. 25.2%; 95% CI], 1.27-1.62; P < 0.01; I2 Z 42%) 10. The CAD EYE system (Fujifilm) is a CADe device supporting both detection (sensitivity > 95%) and characterization of colonic polyps in real time.

To date, artificial intelligence has never been evaluated for CRC screening in patients followed up for LS. The aim of this work is to evaluate the effectiveness of the CAD EYE system in this specific population. To this end, we intend to conduct a randomized, controlled, non-inferiority trial comparing CAD EYE with CE in patients with LS.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pathogenic mutation (path_MLH1, path_MSH2, path_MSH6, path_PMS2, path_EpCAM)
* Male or female of legal age at time of colonoscopy prescription.
* Patient agreeing to participate in the study
* Person affiliated with or benefiting from a social security scheme
* Free, informed and express consent

Exclusion Criteria:

* Patient undergoing total colectomy with ileoanal or ileosigmoid anastomosis
* Patient with a history of Crohn's disease or ulcerative colitis
* Patients with a known allergy or intolerance to polyethylene glycol and ascorbic acid.
* Patients unable to undergo fractionated colonic preparation
* Inadequate colonic preparation: Boston sub-score <2 per segment
* Patient under guardianship or protected person
* Patient who does not understand French or cannot read
* Person not affiliated to a Social Security system.
* Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2026-04-18 (Estimated)

PRIMARY OUTCOMES:
to evaluate the effectiveness of the CAD EYE system in screening for neoplastic lesions in Lynch syndrome. | Through study completion, an average of 2 years
  Comparison of the adenoma detection rate (ADR) between the CAD-EYE group and the indigo carmin chromoendoscopy (CE) group (reference technique).

SECONDARY OUTCOMES:
Detection rates of specific lesions | Through study completion, an average of 2 years
  Mean number of adenomas and serrated lesions per patient
Diagnostic performance of CAD EYE | Through study completion, an average of 2 years
  Comparison of the diagnostic performance of CAD EYE assessed by specificity, negative predictive value and positive predictive value for the characterization (adenoma/hyperplastic) of colonic polyps with the CAD EYE automated detection system. The anatomopathology of polyps was taken as the diagnostic reference.
Rate of resect and discard strategy | Through study completion, an average of 2 years
  Evaluation of the feasibility of a "resect and discard" strategy in Lynch Syndrome. Retrospective analysis comparing CAD-EYE histological prediction vs. endoscopist prediction, using histological report as reference examination (Sensitivity and negative predictive value).
Time of Colonoscopies | Through study completion, an average of 2 years
  Comparison of different procedure times between the 2 groups. Total procedure time will be defined as the time from endoscope insertion to extraction through the anus. Withdrawal time will be defined as the time spent on inspection, from the cecum to extraction of the endoscope through the anus, excluding the time required for polypectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Européen Georges-Pompidou HEGP, Paris, France